CLINICAL TRIAL: NCT00228189
Title: Induction of Specific T Cell Responses in Colorectal Cancer Patients With Liver Metastases Upon Vaccination With Autologous Dendritic Cells Pulsed With CEA-peptide or Electroporated With CEA-RNA: Evaluation of in Vivo Immune Response.
Brief Title: Carcinoembryonic Antigen-loaded Dendritic Cells in Advanced Colorectal Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: C.J.A. Punt, MD, PhD, Radboud University Nijmegen Medical Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 920-03-250; NWO920-03-250
Record Dates: First submitted 2005-09-27; First posted 2005-09-28 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: Dendritic cells; Colorectal cancer; Carcinoembryonic antigen; Vaccine; Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms

ARMS (3):
- A (Active Comparator): Dendritic cells pulsed with CEA-peptide
  Interventions: Biological: CEA-loaded dendritic cell vaccine
- B (Experimental): Dendritic cells electroporated with CEA-mRNA
  Interventions: Biological: CEA-loaded dendritic cell vaccine
- C (Experimental): Dendritic cells pulsed with CEA-peptide, in combination with oxaliplatin/capecitabine
  Interventions: Biological: CEA-loaded dendritic cell vaccine

INTERVENTIONS:
Biological: CEA-loaded dendritic cell vaccine — Carcinoembryonic antigen (either peptide or mRNA) loaded dendritic cells.

SUMMARY:
Dendritic cells (DCs) are the professional antigen-presenting cells of the immune system. As such they are currently used in clinical vaccination protocols in cancer patients. We evaluate the ability of mature DCs pulsed with carcinoembryonic antigen (CEA)-peptide (arm A) or electroporated with CEA-mRNA (arm B) to induce CEA-specific T cell responses in patients with resectable liver metastases from colorectal cancer. To evaluate immune responses, CEA-specific T cell reactivity is monitored in peripheral blood, resected abdominal lymph nodes, tumor tissue and biopsies of vaccination sites and post-treatment DTH skin tests. Patients are vaccinated intradermally and intravenously with CEA-peptide pulsed mature DCs three times prior to resection of liver metastases. In 2007 a side-study has been added (arm C), in which patients with stage III or high-risk stage II colorectal cancer that are amenable for standard adjuvant oxaliplatin/capecitabine therapy are vaccinated with CEApeptide-pulsed DCs. Also in this group, safety and immune responses in peripheral blood and the DTH-skin test are the primary endpoints. Results are compared with the results obtained in arm A.

ELIGIBILITY:
For arm A and B

Inclusion Criteria:

1. Histological documented evidence of colorectal cancer.
2. Primary tumor surgically removed, recurrence(s) in the liver.
3. Planned surgical excision of liver metastases.
4. HLA-A2.1 phenotype according to lymphocyte HLA typing.
5. Expression of CEA on primary tumor.
6. ECOG performance status 0-1, life expectancy > 3 months.
7. Age 18-75 years.
8. WBC > 3.0 x 109/l, lymphocytes > 0.8 x 109/l, platelets > 100 x 109/l, serum creatinine < 150 μmol/l, serum bilirubin < 25 μmol/l.
9. Expected adequacy of follow-up.
10. Written informed consent.

Exclusion Criteria:

1. Clinical signs of extra hepatic metastases, in patients with a clinical suspicion of other metastases diagnostic tests should be performed to exclude this.
2. Prior chemotherapy, immunotherapy, or radiotherapy within three months before planned surgical excision is allowed.
3. A history of myocardial infarction, angina pectoris, cardiac arrhythmias, cerebrovascular accidents, transient ischemic attacks or severe hypertension (exclusion criteria for autologous blood donation)
4. Concomitant use of corticosteroids or other immunosuppressive agents.
5. A history of any second malignancy in the past five years excluding adequately treated basal carcinoma of skin or carcinoma in situ of cervix.
6. Serious concomitant disease, active infections. Specifically, patients with autoimmune disease or organ allografts and patients with a history of HBsAg or HIV are excluded.
7. A known allergy to shell fish.
8. Pregnant or lactating women.

For arm C (side-study)

inclusion criteria:

1. histological proof of colorectal cancer
2. HLA-A0201 positive
3. stage III (T1-4N1-2M0) cancer or high risk stage II (T4 and/or poor differentiation in histology and/or perforation and/or obstruction and/or venous invasion and/or histological analysis of ≤10 lymph nodes)
4. ≤ 8 weeks since surgical resection of primary colorectal tumor
5. Age 18-75 years
6. WHO performance 0-1 (Karnofsky 100-70%)
7. WBC ≥ 3.0x109/l
8. Platelets ≥ 100x109/l
9. Hb ≥ 6 mmol/l
10. Total bilirubin ≤ 2x UNL
11. ASAT and ALAT ≤ 3x UNL
12. Serum creatinine ≤ 1.5 x UNL
13. Expected adequacy of follow-up
14. Signed written informed consent

exclusion criteria

1. A history of second malignancy within the last 5 years. Adequately treated basal carcino¬ma of skin or carcinoma in situ of cervix is acceptable within this period
2. Serious concomitant disease. Autoimmune disease or organ grafts.
3. Other serious concomitant diseases preventing the safe administration of study drugs or likely to interfere with the study assessments.
4. A known allergy to shell fish (contains KLH)
5. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
immunological response against carcinoembryonic antigen and the control protein KLH | During the study
Toxicity | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Prof. dr. C.J.A. Punt, MD,PhD, Principal Investigator — Radboud University Nijmegen Medical Center, dept. of Medical Oncology
Locations (1):
- Radboud University Nijmegen Medical Center, dept. of Medical Oncology, Nijmegen, Netherlands

REFERENCES:
- [Background] Figdor CG, de Vries IJ, Lesterhuis WJ, Melief CJ. Dendritic cell immunotherapy: mapping the way. Nat Med. 2004 May;10(5):475-80. doi: 10.1038/nm1039. PMID 15122249
- [Background] Lesterhuis WJ, Aarntzen EH, De Vries IJ, Schuurhuis DH, Figdor CG, Adema GJ, Punt CJ. Dendritic cell vaccines in melanoma: from promise to proof? Crit Rev Oncol Hematol. 2008 May;66(2):118-34. doi: 10.1016/j.critrevonc.2007.12.007. Epub 2008 Feb 8. PMID 18262431
- [Background] de Vries IJ, Bernsen MR, Lesterhuis WJ, Scharenborg NM, Strijk SP, Gerritsen MJ, Ruiter DJ, Figdor CG, Punt CJ, Adema GJ. Immunomonitoring tumor-specific T cells in delayed-type hypersensitivity skin biopsies after dendritic cell vaccination correlates with clinical outcome. J Clin Oncol. 2005 Aug 20;23(24):5779-87. doi: 10.1200/JCO.2005.06.478. PMID 16110035
- [Result] Lesterhuis WJ, de Vries IJ, Schuurhuis DH, Boullart AC, Jacobs JF, de Boer AJ, Scharenborg NM, Brouwer HM, van de Rakt MW, Figdor CG, Ruers TJ, Adema GJ, Punt CJ. Vaccination of colorectal cancer patients with CEA-loaded dendritic cells: antigen-specific T cell responses in DTH skin tests. Ann Oncol. 2006 Jun;17(6):974-80. doi: 10.1093/annonc/mdl072. Epub 2006 Apr 6. PMID 16600979
- [Derived] Lesterhuis WJ, De Vries IJ, Schreibelt G, Schuurhuis DH, Aarntzen EH, De Boer A, Scharenborg NM, Van De Rakt M, Hesselink EJ, Figdor CG, Adema GJ, Punt CJ. Immunogenicity of dendritic cells pulsed with CEA peptide or transfected with CEA mRNA for vaccination of colorectal cancer patients. Anticancer Res. 2010 Dec;30(12):5091-7. PMID 21187495
- See also: Home page of the Radboud University Nijmegen Medical Center — http://www.umcn.nl
- See also: Website of the tumor immunology department of the Nijmegen Center for Molecular Life Sciences of the Radboud University Nijmegen Medical Center — http://www.ncmls.nl/til/Tumorimmunology.asp